CLINICAL TRIAL: NCT02493803
Title: Impact of Dietary Advice on the Progression of Tooth Wear
Acronym: DAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RJ114/N306
Record Dates: First submitted 2015-05-18; First posted 2015-07-10 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-02

CONDITIONS: Erosive Tooth Wear
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receive detailed dietary advice (Experimental): Half of the participants will be randomly allocated to receive detailed dietary advice
  Interventions: Behavioral: Dietary Advice
- Receive standard of care dietary advice (No Intervention): These patients will receive dietary advice which is the current standard of care

INTERVENTIONS:
Behavioral: Dietary Advice — Detailed dietary advice and planning, complete with dietary information sheets which were developed with a dietitian and a dental psychologist
  Arms: Receive detailed dietary advice

SUMMARY:
The aim of this research is to investigate the impact of dietary advice on the progression of tooth wear over 6 months using a randomised clinical trial design. Participants with severe tooth wear will be recruited. Half of those patients will receive a detailed dietary advice and the other half will be receive standard of care dietary advice. Moulds will be made of their mouths at the original appointment and 6 months later. These moulds will be scanned and superimposed to see if there is any difference in their level of tooth wear

DETAILED DESCRIPTION:
A sample size of 60 patients will be recruited separately from an epidemiology study and written informed consent will be obtained. Patients presenting with moderate to severe tooth wear will be recruited. Those with a Basic Erosive Wear Examination (BEWE) cumulative score greater than or equal to 8 but with at least one score of 3 on the occlusal surfaces of the lower molars or the incisal edge of the upper central incisor. After randomisation, an impression will be taken of the upper and lower teeth using a silicone material. One group will receive one-to-one dietary advice (with dietary information sheets) as the intervention and the other group will not receive any intervention. The silicone impressions will be repeated 6 months later. Impressions will be cast in stone and the occlusal surfaces of the upper or lower molars and the buccal surface of the upper central and lateral incisors will be scanned to monitor tooth wear progression. The two scans of the involved teeth will be superimposed and the level of tooth wear over that time will be calculated.

The investigators aim to see if giving detailed dietary advice will result in less erosive tooth wear.

ELIGIBILITY:
Inclusion Criteria:

1. Severe tooth wear with a BEWE score of 3 on the occlusal surface of the first lower molars or incisal/buccal surface of the upper central incisor.
2. This wear will be as a result of a high acid diet i.e. as at least two dietary acidic challenges a day.
3. Adult 25-70 years old.
4. Minimum of at least 10 occluding tooth pairs (i.e. at least 10 upper teeth which bite against 10 lower teeth) - including the opposing upper molars and lower incisors
5. No anterior crowns/ bridges or implants opposing the lower molars or upper incisors
6. Written consent to the study

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Medical history likely to impact on attendance or mobility
3. Presence of periodontal disease or caries on more than one tooth. BPE score of 2 or above.
4. Unable to speak or understand English
5. Saliva diagnoses (xerostomia- dry mouth)
6. Orthodontic appliances
7. Severe dentine hypersensitivity
8. Restoration of the occlusal or incisal surfaces of upper anterior teeth and first molars.
9. Have factors which could contraindicate their participation, such as any condition requiring the need for antibiotic premedication prior to a dental treatment, a condition requiring the need for long-term antibiotic use, blood thinning medications that prohibit the safe conduct of a dental cleaning or previous use of the weight loss medications.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Loss of tooth height | 6 months
  Models of the teeth taken at 6 month epochs will be scanned using a laser profilometer and superimposed to detect accurately the loss of tooth height that has occurred during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Dental Institute, Guy's Hospital, London, United Kingdom